CLINICAL TRIAL: NCT05494203
Title: Multi-omics Study and Drug Intervention Study of Spondyloarthritis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, XiaobingWang, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: XiaobingWang
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, fecal sample, saliva, Plaque
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spa: Untreated patients meeting the revised AS New York diagnostic criteria or the ASAS classification criteria for axial SpA. Exclusion criteria: ① Patients with rheumatoid arthritis, scleroderma, systemic lupus erythematosus and other diseases of the immune system; ② Patients who have received head and neck radiation therapy; ③ Those who have a history of using antidepressants and parasympathetic stimulants; ④ Known infection with human immunodeficiency virus (HIV) or hepatitis C virus; ⑤ Patients with sarcoidosis or tuberculosis infection. According to the existing ethical approval documents, the patients signed the informed consent.
  Interventions: Diagnostic Test: questionnaire survey
- HC: healthy control. Exclusion criteria: ① Patients with rheumatoid arthritis, scleroderma, systemic lupus erythematosus and other diseases of the immune system; ② Patients who have received head and neck radiation therapy; ③ Those who have a history of using antidepressants and parasympathetic stimulants; ④ Known infection with human immunodeficiency virus (HIV) or hepatitis C virus; ⑤ Patients with sarcoidosis or tuberculosis infection. According to the existing ethical approval documents, the patients signed the informed consent.

INTERVENTIONS:
Diagnostic Test: questionnaire survey — All patients received lifestyle questionnaire, medical history, physical signs, auxiliary examination and laboratory examination results before treatment.
  Groups: spa

SUMMARY:
Spondyloarthritis (SpA) is a type of chronic inflammatory rheumatic disease that mainly affects the spine and peripheral joints, or joints, ligaments and tendons. This disease subtype has the same clinical and immunological features. Further explore the pathogenesis of spondyloarthritis, explore the guiding significance of different imaging examinations for spondyloarthritis, and study the efficacy and mechanism of different drugs for spondyloarthritis.

DETAILED DESCRIPTION:
1. Clinical phenotype research. The clinical phenotype is the symptoms and signs of the disease and its evolution. Through the clinical phenotype research of spondyloarthritis, it is helpful to realize the diagnosis and grading of spondyloarthritis and help to achieve individualization Precise treatment.
2. Transcriptomic research. The key genes and pathways involved in the pathogenesis of spondyloarthritis can be explored through transcriptomic research of spondyloarthritis, which can provide help for early diagnosis and seeking potential treatment methods.
3. Microbiological research. Through the microbiome research on spondyloarthritis, the composition and function of intestinal flora in patients with spondyloarthritis can be deeply analyzed to provide help for diagnosis and treatment.
4. Radiomics research. Through the radiomics research on spondyloarthritis, it is helpful to realize the diagnosis and grading of spondyloarthritis and the evaluation and prediction of treatment.
5. Drug treatment research By studying the therapeutic effects of different drugs in patients with spondyloarthritis, it is helpful to explore the efficacy and mechanism of different drugs on spondyloarthritis, and to achieve precise and individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the revised AS New York diagnostic criteria or ASAS axial SpA classification criteria.

Exclusion Criteria:

* patients with rheumatoid arthritis, scleroderma, systemic lupus erythematosus and other immune system diseases;
* patients who had received head and neck radiotherapy;
* patients with history of antidepressants and parasympathetic stimulants;
* patients known to be infected with human immunodeficiency virus (HIV) or hepatitis C virus;
* patients with sarcoidosis or tuberculosis infection.
* patients with inflammatory bowel disease or uveitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Long-term outcomes after treatment | 1 year
  disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaobing Wang, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No